# REPUBLIC OF Turkiye ANKARA YILDIRIM BEYAZIT UNIVERSITY INSTITUTE OF HEALTH SCIENCES

# EVALUATION OF THE EFFECTIVENESS OF VIRTUAL REALITY APPLICATION DURING CESAREAN DELIVERY UNDER SPINAL ANESTHESIA

INFORMED CONSENT FORM FOR PREGNANT WOMEN IN THE CONTROL GROUP

Ankara- 20.12.2024

## CONTROL GROUP PREGNANT INFORMED CONSENT FORM

#### PLEASE TAKE TIME TO READ THIS DOCUMENT CAREFULLY

You are invited to participate in a research study titled "Evaluation of the Effectiveness of Virtual Reality Application During Cesarean Delivery in Pregnant Women Undergoing Spinal Anesthesia" conducted by Prof. Dr. Sena KAPLAN. Before deciding whether to participate in this study, it is important for you to understand why the research is being conducted and what it will involve. Therefore, it is essential that you read and understand this form. If there is anything unclear or you would like more information, please feel free to ask us.

Participation in this study is completely voluntary. You have the right to refuse participation or to withdraw at any time during the study. Responding to this form will be interpreted as your consent to participate. While answering the questions in the provided forms, please do not feel under any pressure or persuasion. The information obtained from these forms will be used solely for research purposes.

# 1. Information About the Study:

### a. Purpose of the Study:

To evaluate the effectiveness of a virtual reality application during cesarean delivery in pregnant women undergoing spinal anesthesia.

#### Study Content:

Data will be collected using the Personal Information Form, Pregnant Monitoring Form, Spielberger State-Trait Anxiety Inventory, and the Maternal Satisfaction During Delivery Evaluation Scale (Cesarean Delivery). Participants will receive training on virtual reality goggles before cesarean delivery. A pre-test of the virtual reality goggles will be conducted in the patient room before the cesarean. The virtual reality goggles will then be used in the cesarean delivery unit.

[] Scientific research [X] Thesis study

c. Estimated Duration of the Study:

The duration for completing the questionnaires and scales before cesarean delivery is approximately 10 minutes.

d. Expected Number of Participants/Volunteers:

The study aims to include 30 individuals who meet the inclusion criteria.

e. Location(s) of the Study:

Ankara University Health Practice and Research Hospitals, Cebeci Hospital, Department of Obstetrics and Gynecology, Cesarean Delivery Unit.

# 2. Participation Consent:

I have read the above information that should be provided to the participant/volunteer prior to the research. I fully understand the scope and purpose of the study I am invited to participate in, as well as the responsibilities I will undertake voluntarily.

The researcher named below provided me with both written and verbal explanations about the study. I had the opportunity to ask questions and received satisfactory answers. I was also verbally informed about the potential risks and benefits of this study. I understand that I can withdraw from the study at any time and for any reason without facing any negative consequences.

Under these conditions, I voluntarily agree to participate in this study, without any pressure or coercion.

Participant's (In Their Own Handwriting)

| Full Name: |
|----------------------------------------------------------------|
| Signature: |
| (If applicable) For Individuals Under Guardianship or Custody: |
| Guardian's or Custodian's (In Their Own Handwriting) |
| Full Name: |
| Signature: |